CLINICAL TRIAL: NCT00849797
Title: Randomized, Open-Label, 2-Way Crossover, Bioequivalence Study of Oxcarbazepine 600 mg Tablet and Trileptal® Following a 600 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Oxcarbazepine 600 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 50370
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxcarbazepine (Experimental): Oxcarbazepine 600 mg Tablet (test) dosed in first period followed by Trileptal® 600 mg Tablet (reference) dosed in second period
  Interventions: Drug: Oxcarbazepine
- Trileptal® (Active Comparator): Trileptal® 600 mg Tablet (reference) dosed in first period followed by Oxcarbazepine 600 mg Tablet (test) dosed in second period
  Interventions: Drug: Trileptal®

INTERVENTIONS:
Drug: Oxcarbazepine — 600 mg Tablet
  Arms: Oxcarbazepine
Drug: Trileptal® — 600 mg Tablet
  Arms: Trileptal®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of a test formulation of oxcarbazepine tablets and Trileptal® tablets administered as a 1 x 600 mg dose under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Male or female, smoker or non-smoker, 18 years of age and older.
* BMI greater than or equal to 19.0 and less than or equal to 30.0 kg/m2

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses or surgery within 4 weeks of the administration of study medication.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than 14 units of alcohol per [1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of 40% alcohol], or positive alcohol breath test at screening.
* Use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, oxcarbazepine, carbamazepine, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to the administration of the study medication.
* Use of an investigational drug or participation on an investigation study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence or neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 30 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days or
* 301 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned or frozen) within 7 days prior to administration of the study medication.
* History or presence of atreoventricular (AV) block.
* Difficulty fasting or consuming the standard meals.
* Intolerance to venipunctures.
* Clinically significant history of renal, hepatic, or cardiovascular, tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Positive urine pregnancy test at screening.
* Breast-feeding subject.
* Female subjects of child-bearing potential having unprotected sexual intercourse with any non-sterile male partner within 14 days prior to study drug administration. Acceptable methods of contraception:
* Intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration.
* Condom or diaphragm + spermicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxcarbazepine (Test) First: Oxcarbazepine 600 mg Tablet (test) dosed in first period followed by Trileptal® 600 mg Tablet (reference) dosed in second period
- Trileptal® (Reference) First: Trileptal® 600 mg Tablet (reference) dosed in first period followed by Oxcarbazepine 600 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Oxcarbazepine (Test) First | Trileptal® (Reference) First
Started | 60 | 60
Completed | 59 | 59
Not Completed | 1 | 1
Not completed — bad veins | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Washout: One Week
Arm/Group | Oxcarbazepine (Test) First | Trileptal® (Reference) First
Started | 59 | 59
Completed | 59 | 57
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Oxcarbazepine (Test) First | Trileptal® (Reference) First
Started | 59 | 57
Completed | 59 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxcarbazepine (Test) First | Trileptal® (Reference) First | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 56 | 114
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 35 | 33 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 48 | 51 | 99
  American Hispanic | 6 | 7 | 13
  Black | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Oxcarbazepine in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Oxcarbazepine: Oxcarbazepine 600 mg Tablet (test) dosed in either period
- Trileptal®: Trileptal® 600 mg Tablet (reference) dosed in either period
Arm/Group | Oxcarbazepine | Trileptal®
Number analyzed (Participants) | 116 | 116
ng/mL | 3537.63 (1333.09) | 3820.31 (1357.08)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 90.86, 90% CI [85.47 to 96.60] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - Oxcarbazepine
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oxcarbazepine | Trileptal®
Number analyzed (Participants) | 116 | 116
ng*h/mL | 9679.79 (2371.03) | 9772.18 (2350.44)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 98.60, 90% CI [96.59 to 100.66] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant) - Oxcarbazepine
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oxcarbazepine | Trileptal®
Number analyzed (Participants) | 116 | 116
ng*h/mL | 9445.55 (2327.24) | 9539.53 (2293.33)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 98.74, 90% CI [96.71 to 100.80] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

4. Secondary Outcome: Cmax - 10-hydroxy-carbazepine in Plasma
Description: Informational Purposes Only
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trileptal: Trileptal® 600 mg Tablet (reference) dosed in either period
Arm/Group | Oxcarbazepine | Trileptal
Number analyzed (Participants) | 116 | 116
ng/mL | 9349.83 (1739.68) | 9517.52 (2034.08)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 98.50, 90% CI [95.66 to 100.48] — Results presented for informational purposes only; metabolite not subjected to bioequivalence criteria

5. Secondary Outcome: AUC0-inf - 10-Hydroxy-Carbazepine Metabolite
Description: Informational Purposes Only
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oxcarbazepine | Trileptal®
Number analyzed (Participants) | 116 | 116
ng*h/mL | 197864.34 (47069.89) | 196607.20 (43337.72)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 100.29, 90% CI [98.96 to 101.64] — Results presented for informational purposes only, metabolite not subjected to bioequivalence criteria

6. Secondary Outcome: AUC0-t - 10-Hydroxy-Carbazepine Metabolite
Description: Informational Purposes Only
Time Frame: Blood samples collected over 48 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oxcarbazepine | Trileptal®
Number analyzed (Participants) | 116 | 116
ng*h/mL | 179002.40 (39157.51) | 177979.76 (35506.55)
Statistical Analysis 1: Comparison: Oxcarbazepine vs Trileptal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 100.08, 90% CI [98.91 to 101.27] — Results presented for informational purposes only; metabolite not subjected to bioequivalence criteria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.